CLINICAL TRIAL: NCT05202548
Title: Immunology Dysregulation in Lymphadenitis Tuberculosis : An Observational Study Using Patient' Block Paraffins 2019 Until 2021
Status: Completed | Type: Observational
Sponsor: Universitas Katolik Widya Mandala Surabaya (Other)
Collaborators: Indonesia's Ministry of Research and Technology (Ristekdikti/BRIN) (Unknown)
Responsible Party: Principal Investigator, Bernadette Dian Novita, MD.,PhD, MD.,PhD, Universitas Katolik Widya Mandala Surabaya
Other Study IDs: 002/AMD-SP2H/LT-MULTIPDPK/LL7
Record Dates: First submitted 2022-01-08; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Lymphadenitis, Tuberculous; Immune Defect
Keywords: Lymphadenitis tuberculosis; C-C Chemokines receptor - 2 (CCR-2); C-C Chemokines ligand - 5 (CCL-5); Cytokines inflammatory
MeSH Terms: conditions — Tuberculosis, Lymph Node

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lymphadenitis TB: The group study was blocked paraffin from lymphadenitis tuberculosis patient that already confirmed diagnosis histopathological anatomy (PA histopathology)
  Interventions: Other: Immuno-histochemical staining

INTERVENTIONS:
Other: Immuno-histochemical staining — blocked paraffin that suit with inclusion and exclusion criteria proceed with immuno-histochemical staining to define immune dysregulation in lymphadenitis TB

SUMMARY:
Mycobacterium tuberculosis (M. tuberculosis) infection is still a problem that cannot be overcome in Indonesia. In 2018 the number of tuberculosis (TB) sufferers in Indonesia reached more than 850/100,000 population, an increase around 20% from the previous year's incidence. One of the highest number of cases is in East Java Province, which is 38% of the total number of new TB cases in Indonesia.

Extrapulmonary tuberculosis (EPTB) according to WHO classification criteria is an M. tuberculosis infection that occurs in tissues and organs outside the lung parenchyma. The incidence rate in Indonesia reaches 1-5% of the incidence of TB thus EPTB may often be forgotten. However, the diagnosis, therapy and monitoring post treatment in EPTB remains difficult to do.

The focus of this research is tuberculous lymphadenitis (TB), due to 50% of EPTB cases in Indonesia was lymphadenitis TB. The risk factors for EPTB are immunocompromised conditions, such as HIV infection or comorbid conditions such as chronic kidney disease (CKD) and diabetes mellitus, but the mechanism of EPTB homing is still unclear. The mechanism of EPTB homing, especially TB lymphadenitis, really needs to be known for the development of diagnostics and therapy as well as preventing the occurrence of TB lymphadenitis.

The importance of this research is to obtain compounds from the human immune response that can be developed as diagnostic markers and therapeutic targets for tuberculosis infection, especially TB lymphadenitis. Activated macrophages containing M. tuberculosis are carried by lymph flow to lymph nodes, where there is deposition of antigen-antibody complexes which then activate CC Chemokine Receptor-2 (CCR2) on lymphocytes, which are the primary receptors for Chemokine (CC motif) ligands ( CCL)-8 and CCL5, proteins expressed on macrophages containing M. tuberculosis. Activation of CCR2 increases the production of IL-10(10). IL-10 has been responsible for decreasing the secretion of TNF-, IFN-γ, and IL-1β (11). IFN-γ affects the process of M. tuberculosis elimination and the success of TB therapy, so that IL-10 is responsible for the failure of macrophages to eliminate M. tuberculosis. IL-10 also binds to Signal Transducer and Activator of Transcription 3 (STAT3) and STAT3 increases the release of Suppressor of Cytokine Signaling 3 (SOCS3). SOCS3 interferes with IFN-γ signaling for CCR2 recognition of M. tuberculosis-containing macrophages. On the other hand, the mechanism of T lymphocytes and macrophages that activate pro-inflammatory mediators (TNF-, IFN-γ, and IL-1β) and the association of IL-10 activation on STAT3, SOCS3 and CCR2 expression in the incidence of EPTB, especially TB lymphadenitis without TB infection remains unknown.

DETAILED DESCRIPTION:
Mycobacterium tuberculosis (M. tuberculosis) infection is still a problem that cannot be overcome in Indonesia. In 2018 the number of tuberculosis (TB) sufferers in Indonesia reached more than 850/100,000 population, an increase around 20% from the previous year's incidence. One of the highest number of cases is in East Java Province, which is 38% of the total number of new TB cases in Indonesia.

Extrapulmonary tuberculosis (EPTB) according to WHO classification criteria is an M. tuberculosis infection that occurs in tissues and organs outside the lung parenchyma. The incidence rate in Indonesia reaches 1-5% of the incidence of TB thus EPTB may often be forgotten. However, the diagnosis, therapy and monitoring post treatment in EPTB remains difficult to do.

The focus of this research is tuberculous lymphadenitis (TB), due to 50% of EPTB cases in Indonesia was lymphadenitis TB. The risk factors for EPTB are immunocompromised conditions, such as HIV infection or comorbid conditions such as chronic kidney disease (CKD) and diabetes mellitus, but the mechanism of EPTB homing is still unclear. The mechanism of EPTB homing, especially TB lymphadenitis, really needs to be known for the development of diagnostics and therapy as well as preventing the occurrence of TB lymphadenitis.

The importance of this research is to obtain compounds from the human immune response that can be developed as diagnostic markers and therapeutic targets for tuberculosis infection, especially TB lymphadenitis. Activated macrophages containing M. tuberculosis are carried by lymph flow to lymph nodes, where there is deposition of antigen-antibody complexes which then activate CC Chemokine Receptor-2 (CCR2) on lymphocytes, which are the primary receptors for Chemokine (CC motif) ligands ( CCL)-8 and CCL5, proteins expressed on macrophages containing M. tuberculosis. Activation of CCR2 increases the production of IL-10(10). IL-10 has been responsible for decreasing the secretion of TNF-, IFN-γ, and IL-1β (11). IFN-γ affects the process of M. tuberculosis elimination and the success of TB therapy, so that IL-10 is responsible for the failure of macrophages to eliminate M. tuberculosis. IL-10 also binds to Signal Transducer and Activator of Transcription 3 (STAT3) and STAT3 increases the release of Suppressor of Cytokine Signaling 3 (SOCS3). SOCS3 interferes with IFN-γ signaling for CCR2 recognition of M. tuberculosis-containing macrophages. On the other hand, the mechanism of T lymphocytes and macrophages that activate pro-inflammatory mediators (TNF-, IFN-γ, and IL-1β) and the association of IL-10 activation on STAT3, SOCS3 and CCR2 expression in the incidence of EPTB, especially TB lymphadenitis without TB infection remains unknown.

In this study, Lymphadenitis TB paraffin blocks from patients were collected and screened for immunological responses that TB patients have potential as targets for diagnosis and therapy. The paraffin block samples came from the Anatomical Pathology Laboratory of St. Catholic Hospital. Vincentius A Paulo (RKZ) Surabaya. Existing samples were taken and performed immuno-histochemical (IHC) to define theimmune dysregulation in TB lymphadenitis.

ELIGIBILITY:
Inclusion Criteria:

* Lymphadenitis TB blocked paraffin that already confirmed by the Pathologist and MPT64 staining

Exclusion Criteria:

* broken blocked paraffin due to the storage process

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population in this study was blocked paraffin that diagnosed with lymphadenitis TB by pathologist and confirmed with MPT64 staining
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
IHC slides | 15 November 2021
  Histopathology slides stained by immuno-histochemical substrates

CONTACTS AND LOCATIONS:
Locations (1):
- Vincentius A Paulo Surabaya Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
Study protocol share

REFERENCES:
- [Derived] Novita BD, Tjahjono Y, Wijaya S, Theodora I, Erwin F, Halim SW, Hendrawan B, Jaya DK, Tahalele PL. Characterization of chemokine and cytokine expression pattern in tuberculous lymphadenitis patient. Front Immunol. 2022 Nov 10;13:983269. doi: 10.3389/fimmu.2022.983269. eCollection 2022. PMID 36439164